CLINICAL TRIAL: NCT06771427
Title: Systemic Proteomic Analysis of Plasma Exosomes to Explore the Immunomodulation Reflected to Sjogren's Syndrome and Dry Eye Syndrome
Brief Title: Exosomes Proteomic for Sjogren's Syndrome and Dry Eye Syndrome
Status: Recruiting | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ching-Mao Chang, Director of Division of Integrative Medicine, Center for Traditional Medicine, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2024-07-018BC
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye Syndrome (DES); Sjogren's Syndrome; Xerophthalmia
Keywords: Dry eye syndrome; Sjögren's syndrome; Xerophthalmia; Chinese herbal tea; Nourishing Yin and Moistening Dryness; Exosome; GB20; BL2; proteomics
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome; Xerophthalmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — This study will analyze remaining samples from TBDESJS and ACUDES participants, aiming to extend the analysis to 80 DES and 110 SJS participants, and 30 NHC, and then we identified the 40 DES participants and 60 SJS participants who exhibited the most significant therapeutic improvement pre- and post-treatment, alongside 30 healthy control subjects. The study will systematically analyze exosome-miRNA and transcriptome to investigate the possible mechanisms by which Chinese herbal tea bags and acupuncture alleviate dryness symptoms in the mouth and eyes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Group GB20: Group GB20 will received acupuncture at acupoint GB20 twice a week 8 weeks for efficacy evaluation. And we could use the proteomic, exosome-proteomic, , exosome-miRNA, transcriptome, oral microbiota, Schirmer's test, Tear breakup time, 6-GSI, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Other: acupuncture GB20 or GB20 plus BL2
- Group GB20 plus BL2: Group GB20 plus BL2 will received acupuncture at acupoint GB20 plus BL2 twice a week 8 weeks for efficacy evaluation. And we could use the proteomic, exosome-proteomic, exosome-miRNA, transcriptome, oral microbiota, Schirmer's test, Tear breakup time, 6-GSI, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Other: acupuncture GB20 or GB20 plus BL2
- non AIDDES Healthy Controls (NHC): ACUDES: Healthy control group will not received any treatment. And we could use the proteomic, exosome-proteomic, exosome-miRNA, transcriptome, oral microbiota, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability to find the difference with the comparison between the dry eye syndrome and healthy control.
  TBDESJS: Non DES SJS Healthy Controls (NHC) will received Chinese herbal tea TBDESJS 8 weeks on Nourishing Yin and Moistening Dryness the ocular dryness evaluation. And we could use the Schirmer's test, Tear breakup time, Ocular Surface Disease Index (OSDI), EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI), Pittsburgh Sleep Quality Index (PSQI), Ford Insomnia Response to Stress Test (FIRST), cytokine markers, Whole-genome genotyping, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Other: acupuncture GB20 or GB20 plus BL2; Drug: Chinese herbal tea TBDESJS
- Waiting list: Group Waiting list will not received any treatment. at acupoint GB20 plus BL2 twice a week 8 weeks for efficacy evaluation. And we could use the proteomic, exosome-proteomic, exosome-miRNA, transcriptome, oral microbiota, Schirmer's test, Tear breakup time, 6-GSI, OSDI, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Drug: Chinese herbal tea TBDESJS
- Dry eye syndrome (DES): Dry eye syndrome (DES) will received Chinese herbal tea TBDESJS 8 weeks on Nourishing Yin and Moistening Dryness the ocular dryness evaluation. And we could use the proteomic, exosome-proteomic, exosome-miRNA, transcriptome, Schirmer's test, Tear breakup time, Ocular Surface Disease Index (OSDI), EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI), Pittsburgh Sleep Quality Index (PSQI), Ford Insomnia Response to Stress Test (FIRST), cytokine markers, Whole-genome genotyping, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Drug: Chinese herbal tea TBDESJS
- Sjögren's syndrome (SJS): Sjögren's syndrome (SJS) will received Chinese herbal tea TBDESJS 8 weeks on Nourishing Yin and Moistening Dryness the ocular dryness evaluation. And we could use the proteomic, exosome-proteomic, exosome-miRNA, transcriptome, Schirmer's test, Tear breakup time, Ocular Surface Disease Index (OSDI), EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI), Pittsburgh Sleep Quality Index (PSQI), Ford Insomnia Response to Stress Test (FIRST), cytokine markers, Whole-genome genotyping, TCM pattern, Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, and TCM heart rate variability for this purpose.
  Interventions: Drug: Chinese herbal tea TBDESJS

INTERVENTIONS:
Other: acupuncture GB20 or GB20 plus BL2 — acupuncture at acupoint GB20 or GB20 plus BL2 twice a week 8 weeks for efficacy evaluation.
  Groups: Group GB20; Group GB20 plus BL2; non AIDDES Healthy Controls (NHC)
Drug: Chinese herbal tea TBDESJS — Chinese herbal tea TBDESJS 8 weeks on Nourishing Yin and Moistening Dryness the ocular dryness evaluation.
  Groups: Dry eye syndrome (DES); Sjögren's syndrome (SJS); Waiting list; non AIDDES Healthy Controls (NHC)

SUMMARY:
By analyzing the differential proteins in exosomes, this study aims to understand the pathological mechanisms of SJS and DES, identify potential diagnostic and therapeutic methods, and advance the diagnosis and treatment of these diseases.

DETAILED DESCRIPTION:
Background: A 2015 survey in Taiwan revealed that the prevalence of Dry Eye Syndrome (DES) is 4.87%, with 4.8% of these cases likely to develop into Sjögren's Syndrome (SJS). An American study indicated that 11.6% of DES cases could be diagnosed as SJS, and SJS patients showed significantly more severe conjunctival and corneal staining, Schirmer's test results, clinical symptoms, anti-nuclear antibody, and rheumatoid factor compared to non-SJS patients. Various autoimmune diseases (such as SJS, SLE, RA, SSc, AS, etc.) also affect the severity of dry eye symptoms. Recent studies have employed exosome proteomics to investigate cell-to-cell communication, molecular mechanisms of diseases, and the development of new diagnostic markers and therapeutic targets. While these studies have significant research value for understanding disease mechanisms, diagnosis, and treatment, few have specifically focused on the impact of exosome proteomics in SJS and DES.

Objective: By analyzing the differential proteins in exosomes, this study aims to understand the pathological mechanisms of SJS and DES, identify potential diagnostic and therapeutic methods, and advance the diagnosis and treatment of these diseases.

Methods: This study will develope on previous research projects conducted at Taipei Veterans General Hospital (TBDESJS，V112C-190) and the National Science and Technology Council (ACUDES). TBDESJS focused on evaluating the use of a herbal tea TBDESJS for relieving dry eye and mouth symptoms in DES and SJS patients, and ACUDES explored the immediate and long-term effects of acupuncture on treating dry eye and mouth symptoms in DES and SJS patients by using the GB20 (Fengchi) and BL2 (Zanzhu) acupuncture points.

1. TBDESJS Study: Included 30 DES patients, 60 SJS patients, and 10 healthy controls (NHC) to evaluate the efficacy of the Traditional Chinese Medicine (TCM) herbal tea in improving dry eye and mouth symptoms.
2. ACUDES Study: Included 50 DES patients, 50 SJS patients, and 20 NHC to evaluate the efficacy of acupuncture GB20 and BL2 in improving dry eye and mouth symptoms.

The study will further analyze the remaining samples from these two projects with consent from the participants (45 SJS, 28 DES, and 10 NHC from TBDESJS; 47 SJS, 40 DES, and 20 NHC from ACUDES). In total, 92 SJS, 68 DES, and 30 NHC participants will be included. We will select 40 participants with significant therapeutic improvement from the ACUDES study and 40 from the TBDESJS study for pre- and post-treatment comparison, along with 20 NHC participants, total 100 subjects and 180 person-times.

Additionally, we will perform comprehensive cross-analyses incorporating whole-genome genotyping, cytokines, Schirmer's test, tear breakup time, TCM constitution scale, OSDI, ESSPRI, PSQI, FIRST, TCM pulse diagnosis, TCM tongue diagnosis, and TCM heart rate variability measurements. This will help us understand the potential pathways by which the TBDESJS and ACUDESJS regulate immunity, aiming for future clinical applications in SJS and DES patients, ultimately achieving the goal of Holistic Health Care.

Expected Outcomes:

1. Purify exosomes from the plasma of SJS and DES patients, identify differential proteins between healthy individuals and patients, and investigate the roles of these proteins in immune cell regulation and their potential as diagnostic tools.
2. Analyze the differential proteins in plasma exosomes of SJS and DES patients before and after treatment with the TBDESJS and ACUDES to explore their therapeutic mechanisms.
3. Explore the possible pharmacological mechanisms of the TBDESJS and ACUDES.

ELIGIBILITY:
Dry eye syndrome

Inclusion Criteria: aged between 20 and 75 years Schirmer's test less than 10 mm/5 min Exclusion Criteria: Pregnancy With eye inflammation or infectious eye disease Accepted operation of eye Sjögren's syndrome

Inclusion Criteria: primary or secondary SS aged between 20 and 75 years fulfilled the 2002 American-European Consensus Criteria for SS (AECG) had no abnormal findings of immune, liver, kidney, or blood function evaluations.

Exclusion Criteria: a history of alcohol abuse, diabetes mellitus, or major life-threatening condition pregnancy or breastfeeding steroid pulse therapy within three months prior to the commencement of our study.

non AIDDES Healthy Controls

Inclusion Criteria: aged between 20 and 75 years without any Chronic disease Exclusion Criteria: any Sjögren's syndrome or Dry eye syndrome.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dry Eye Syndrome (DES):
  Participants diagnosed with Dry Eye Syndrome, characterized by symptoms such as ocular discomfort, dryness, and visual disturbances.
  Sjögren's Syndrome (SS):Patients diagnosed with Sjögren's Syndrome, an autoimmune disorder marked by dry eyes and mouth, often accompanied by systemic manifestations.
  non AIDDES Healthy Controls (NHC): Healthy individuals without any history of dry eye symptoms or autoimmune diseases, serving as a control group.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Schirmer's test | 8 weeks
  Dry eye syndrome (DES) and Sjögren's syndrome (SJS) take the Schirmer's test.
Ocular Surface Disease Index (OSDI) | 8 weeks
  Dry eye syndrome (DES) and Sjögren's syndrome (SJS) take the OSDI(Ocular Surface Disease Index).

SECONDARY OUTCOMES:
TCM pattern | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM pattern to differentiate the 9 types of TCM constitutions.
TCM tongue diagnosis | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM tongue diagnosis with camera photo to differentiate the TCM tongue feature factors about Tongue body, Tongue Coating, Red spot, Tooth marks, and Ecchymosis. TCM tongue feature factors would present the status of inflammation, blood stasis, heat, dampness with TCM theory.
TCM pulse diagnosis | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM pulse diagnosis with blood pressure monitors to differentiate the TCM pulse feature factors about Floating, Deep, Slow, Rapid, Deficient, Excessive, Slippery, Rough, String-like, Soggy, Fine, Weak. TCM tongue feature factors would present the status of inflammation, blood stasis, heat, dampness with TCM theory.
TCM heart rate variability | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the TCM heart rate variability.
Whole-genome genotyping(TWBv2.0) | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls (NHC) take the Whole-genome genotyping (TWBv2.0).
Cytokine markers | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the cytokine markers (IL-17, MMP-9, BAFF, BCMA) analysis.
Pittsburgh Sleep Quality Index | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the Pittsburgh Sleep Quality Index
Ford Insomnia Response to Stress Test | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the Ford Insomnia Response to Stress Test.
EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | 8 weeks
  Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC) take the EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI)
Tear breakup time (TBUT) | 8 weeks
  Tear breakup time (TBUT) is a clinical test used to assess for evaporative dry eye disease.
Exosome-miRNA, transcriptome | 8 weeks
  exosome-miRNA, transcriptome can be used to assess for Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC)
Proteomic, Exosome-proteomic | 8 weeks
  Proteomic, Exosome-proteomiccan be used to assess for Dry eye syndrome (DES), Sjögren's syndrome (SJS), and on DES SJS Healthy Controls, NHC)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Mao Chang, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Ching-Mao, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, we have not determined the specifics of IPD sharing. The decision will be based on further considerations, including data availability, privacy concerns, compliance with ethical standards, and potential collaborations with other researchers.

REFERENCES:
- [Background] Lin HC, Yen CM, Chen WS, Hsu CC, Kung YY, Wu JH, Su YT, Chen KF, Chen HY, Lien CM, Wang MJ, Chang CM. Unveiling the age-related dynamics in Sjogren's syndrome: Insights from heart rate variability and autonomic function. Int J Rheum Dis. 2024 Mar;27(3):e15088. doi: 10.1111/1756-185X.15088. PMID 38454192
- [Background] Yen CM, Lin HC, Chen WS, Hsu CC, Liaw CC, Kung YY, Ma CP, Chen HY, Su YT, Chang CM. Evaluation of traditional Chinese medicine tea bag TBDESJS in patients with Sjogren's syndrome and dry eye syndrome: A phase II pilot study. Int J Rheum Dis. 2024 Nov;27(11):e15398. doi: 10.1111/1756-185X.15398. PMID 39473287